CLINICAL TRIAL: NCT04265040
Title: TranslatiOnal Registry for CardiomyopatHies (TORCH) - Plus as Part of the German Centre for Cardiovascular Research (DZHK)
Brief Title: DZHK TORCH-Plus is a Registry for Patients With Cardiomyopathies and Serves as Source for Cardiovascular Research Studies
Acronym: TORCH-Plus
Status: Recruiting | Type: Observational
Sponsor: University Hospital Heidelberg (Other)
Collaborators: University Medicine Greifswald (Other); Charite University, Berlin, Germany (Other); German Heart Center (Other); University of Mannheim (Other); University Hospital Schleswig-Holstein (Other); Medical University of Hannover (Other); Goethe University (Other); Universitätsklinikum Hamburg-Eppendorf (Other); University Medical Center Mainz (Other); University Medical Center Goettingen (Other); Deutsches Herzzentrum Muenchen (Other); Technical University of Munich (Other); University Hospital Munich (Other); Kerckhoff Klinik (Other)
Responsible Party: Principal Investigator, Benjamin Meder, Deputy Director - Clinic of Cardiology, Angiology and Pneumology, University Hospital Heidelberg
Other Study IDs: TORCH-Plus DZHK21
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Non-ischemic Cardiomyopathy; DCM - Dilated Cardiomyopathy; HCM - Hypertrophic Cardiomyopathy; HOCM - Hypertrophic Obstructive Cardiomyopathy; Arrhythmogenic Right Ventricular Cardiomyopathy; Left Ventricular Noncompaction Cardiomyopathy; Amyloidosis; Inflammatory Cardiomyopathy
Keywords: Cardiomyopathies, registry, data, biomaterial, genetics
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathy, Hypertrophic; Arrhythmogenic Right Ventricular Dysplasia; Amyloidosis; Cardiomyopathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The DZHK TranslatiOnal Registry for CardiomyopatHies (DZHK TORCH) represents a unique resource of clinical data and high quality biological samples to enable innovative clinical and molecular studies on cardiomyopathies (CMP). As a multi-center German cardiomyopathy registry, TORCH has been prospectively admitting patients since December 2014. 2,300 patients were recruited as planned. Taken together, patient data showed that the prevalence of these diseases is much higher in men than in women, atrial fibrillation is common in all forms of CMPs as well as rare forms of disease indicate a higher risk and higher morbidity.

This DZHK TORCH register is now to be expanded with a second phase (DZHK TORCH-Plus). The second phase DZHK TORCH-Plus consists of 4 main modules: 1. "Clinical phenotyping, follow-up & biosampling" 2. "Genomics", 3. "Inflammation" and 4. "Biomarker". The central aims are 1) to significantly increase the number of probands (n = 4340) in order to better address the different types of CMPs, especially patients with rare CMP forms such as LVNC and ARVC or with probably molecularly explainable cardiomyopathies (familial DCM), 2) to prolong the longitudinal with a further follow-up to achieve sufficient events and thereby derive clinical recommendations for risk assessment, 3) to increase the number of probands with state-of-the-art phenotyping, 4) to pinpoint the effect of myocardial inflammation, fibrosis, gender and to determine or predict genotypes based for outcome, 5) to validate novel biomarkers developed in other DZHK studies, and 6) to foster active cooperation with international CMP registries and partners from industry.

ELIGIBILITY:
Inclusion Criteria:

* Non-ischemic structural cardiomyopathies
* Age ≥ 18 or ≤ 80 years
* The patient is able to understand the declaration of consent and to sign it dated
* At least one of the following diagnoses depending on the specific TORCH-

Plus inclusion / exclusion - SOP:

Dilated Cardiomyopathy (DCM)

* family / genetic
* inflammatory / persistent myocarditis
* idiopathic (after exclusion secondary cause)
* left sided systolic dysfunction (EF ≤ 45%)

Left ventricular hypertrophy

* sarcomere hypertrophic cardiomoypathia (HCM, HOCM)
* amyloid (AL: light chains, TTR: transthyretin, wild type)

Left ventricular non-compaction cardiomyopathy (LVNC)

Arrhythmogenic right ventricular cardiomyopathy (ARVC / D)

Exclusion Criteria:

The following exclusion criteria have been defined and must be taken from the TORCH-Plus specific inclusion / exclusion - SOP in detail:

* Age: <18 years or> 80 years
* Patient has other (cardiac) previous illnesses:

  * uncontrollable arterial hypertension
  * primary pulmonary arterial hypertension
  * radiation therapy in the chest area
  * addiction (drug or alcohol abuse)
  * life expectancy <1 year due to non-cardiological pre-existing conditions
  * significant heart valve disease
  * ischemic diseases and severe congenital heart diseases (including VSD, Fallot tetralogy, Ebstein anomaly)
  * chemotoxic cardiomyopathy
  * condition after myocarditis
  * combination of several traditional risk factors (e.g. hypertension and diabetes mellitus)
  * advanced chronic non-cardiac disease (e.g. chronic hepatitis or HIV)
  * Tachymyopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 2040 (Estimated)
Dates: Start 2020-08-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
all-cause mortality | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Heidelberg - Clinic of Cardiology, Angiology and Pneumology, Heidelberg, Baden-Wurttemberg, Germany